CLINICAL TRIAL: NCT04578886
Title: The Effect of Guanfacine on Delirium in Critically Ill Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Andrew Barker, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Guanfacine for Delirium
Record Dates: First submitted 2020-09-18; First posted 2020-10-08 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Delirium
Keywords: Delirium; Critically Ill; Guanfacine
MeSH Terms: conditions — Delirium; Critical Illness | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo, lactulose monohydrate, encapsulated, once nightly at 2100, for up to 14 day study duration or otherwise indicated by study protocol.
  Interventions: Drug: Placebo
- Guanfacine (Experimental): Guanfacine immediate-release, 2mg dose, over-encapsulated tablet, once nightly at 2100, for up to 14 day study duration or otherwise indicated by study protocol.
  Interventions: Drug: Guanfacine

INTERVENTIONS:
Drug: Guanfacine — Guanfacine 2 mg administered at 21:00 for up to 14 days or otherwise indicated by study protocol.
  Arms: Guanfacine
Drug: Placebo — Placebo, administered at 2100 for up to 14 days or otherwise indicated by study protocol.
  Arms: Placebo

SUMMARY:
Delirium in patients in the intensive care unit (ICU) is a common problem associated with increased mortality and morbidity, including increased hospital and ICU length of stay, greater hospital cost, increased ventilator days, and long-term cognitive disability. Various pharmacologic agents including dopamine antagonists, acetylcholinesterase inhibitors, melatonin, antipsychotics, alpha-2 agonists, and glutamate antagonists are used for treatment of delirium in the ICU despite the lack of clear evidence of efficacy.Since there is no evidence-based pharmacologic treatment of ICU delirium, current therapy is focused on non-pharmacologic prevention techniques and pharmacologic agents are used once delirium is established. Guanfacine, an alpha-2 agonist, has been identified as a potential medication that may be of benefit in the treatment of delirium. The purpose of this study to investigate the effects of guanfacine versus placebo on delirium in critically ill patients admitted to the ICU and to determine whether guanfacine along with standard of care reduces the duration of delirium, compared to standard of care alone.

DETAILED DESCRIPTION:
Delirium is a common problem in critically ill patients with a reported prevalence in the ICU ranging from 11% to 83%. Delirium has been associated with worse clinical outcomes including increased days on mechanical ventilation, length of hospital stay, cost of care, self-removal of important devices (endotracheal tubes, central venous catheters), use of physical restraint, long-term cognitive impairment, readmission, and mortality. The etiology of delirium is multifactorial, and risk factors include advanced age, substance abuse, metabolic derangements, and sleep disturbances.

Unfortunately, evidence-based strategies for treatment of ICU delirium do not exist. Even with the lack of strong evidence, both non-pharmacologic and pharmacologic therapies are used as standard care in clinical practice. Non-pharmacologic strategies considered as standard care include removal of causative factors, sleep maintenance, reorientation during the day, early mobilization activities, timely removal of catheters and physical restraints, and use of a scheduled pain management protocol. In combination with these non-pharmacologic strategies, ICU patients are treated with pharmacologic agents to render the patient safe and manageable and to promote sleep and normal circadian cycle. Despite lack of an FDA approved drug for treating delirium and clear-cut efficacy of any drug, various pharmacologic agents standardly used to treat delirium in the ICU include dopamine antagonists, acetylcholinesterase inhibitors, melatonin, antipsychotics, alpha-2 agonists, and glutamate antagonists. Antipsychotics, such as haloperidol, have been most commonly used. However, the effectiveness of routinely using antipsychotics in managing delirium has been questioned given the potential for adverse effects, medication interactions, and unproven benefit. Haloperidol can cause serious side effects including Q-T prolongation, sedation, and extrapyramidal symptoms. For this reason the use of haloperidol is less than ideal in the elderly patient population. Recent studies have looked at the perioperative use of dexmedetomidine in mechanically ventilated patients experiencing hyperactive delirium. Dexmedetomidine is a centrally-acting alpha 2 adrenergic receptor (α2-AR) agonist that generally quiets noradrenergic activity, producing sedative, analgesic and antihypertensive effects. When compared to haloperidol, patients receiving dexmedetomidine have fewer ventilation days, shorter ICU length of stay, less need for tracheostomy, and quicker resolution of delirium symptoms. Unfortunately, dexmedetomidine is expensive and delivered as an intravenous infusion.

Guanfacine, an alpha-2A antihypertensive agent with a safe pharmacodynamic profile, has also been reported as treatment of ICU delirium. It has found use as an adjunct therapy in the management of Attention Deficit Hyperactivity Disorder (ADHD). Compared to dexmedetomidine, guanfacine is a pure alpha-2A agonist with higher selectivity for the dorsolateral PFC structures leading to improved neuronal function by enhancing short-term memory. Noting a similarity between the inattention and hyperactivity of emergence and ADHD itself, clinicians have started using guanfacine to manage young, healthy males who were commonly at risk for emergence delirium after anesthesia. In this context, the drug has gained popularity for its off label use perioperatively in a wide variety of patients with anxiety issues, known or predicted to have potential for combative or difficult emergence.

Compared to dexmedetomidine, guanfacine may have a more unique and specific mechanism of behavior modification that could be beneficial as a treatment in delirium. Furthermore, oral guanfacine is cheaper and easier to use, with the ability to continue it outside the ICU. From a pharmacokinetic standpoint, guanfacine is absorbed with peak onset over 1-4 hour and has a half-life of 16 hours. The long half-life allows once-daily dosing before sleep. Maximal drug levels at night promote sleep, with some drug remaining during the day to provide a lesser degree of sedation. Outpatient studies have detected a ceiling effect on the antihypertensive effect of guanfacine, wherein doses of 1 mg, 2 mg, or 3 mg all have the same effect on blood pressure. This implies that up-titrating the guanfacine dose beyond 1 mg daily might increase sedative/hypnotic effects, without increasing hemodynamic instability. Maldonado et al at Stanford has utilized guanfacine for delirious/withdrawing patients (0.5-3 mg total daily dose). A recent case report by Dr. Habib Srour and colleagues described successful use of guanfacine (1 mg q12hr) to control refractory agitation in an ICU patient with a history of opioid misuse.

The investigators propose to perform a pilot trial to evaluate protocol adherence, estimate recruitment rates, and evaluate the safety and efficacy of guanfacine with standard care, compared to standard care alone, on delirium in ICU patients. Before testing other drugs compared with guanfacine, evidence needs to be collected to investigate if guanfacine is more effective than placebo in treating delirium in ICU patients. The control intervention is therefore chosen to be placebo along with standard or usual care. Given the literature and our own experience with the drug for ICU delirium, the investigators plan to use a dose of 2 mg nightly for efficacy and minimization of side effects. The investigators will withhold guanfacine or placebo if a patient does not have delirium for four consecutive assessments or for safety reasons. The investigators will permanently discontinue guanfacine or placebo for any life-threatening, serious adverse event that was related to the intervention. The trial drug or placebo will be discontinued after the 14-day intervention period or at ICU discharge, whichever occurs first.

ELIGIBILITY:
Inclusion criteria

* Patients admitted to the UAB hospital Surgical Intensive Care Unit (SICU)
* 18 years of age or older
* Expected total ICU length of stay of 72 hours or more per treating physician
* Diagnosed with delirium based on CAM-ICU assessment (see attached CAM-ICU assessment form)

Exclusion Criteria

* Patients younger than 18 years old
* Expected discharge from ICU within 72 hours of admission
* Expected or inevitable death with 48 hours of enrollment
* Pregnancy or breast feeding
* Non-English speaking
* Patients unable to be assessed by CAM-ICU due to neurologic illness
* Altered consciousness unable to participate in CAM-ICU assessment
* Patients with previous diagnosis of chronic, acute, subacute neurologic disease, or neurodegenerative disease
* Mental illness and/or psychosis
* Acute alcohol withdrawal
* No enteral route available for administration
* Treating physician refusal of enrollment based on severe hypotension (defined as requiring a vasopressor for longer than 24 hours) or bradycardia (Hr<50 bpm) at the time of screening
* Hepatic encephalopathy
* Blind or Hearing impaired
* Taking Guanfacine, for any reason
* On CYP3A inhibitor such as azole antifungals or clarithromycin
* On CYP3A inducers such as phenytoin or rifampin
* Severe xerostomia
* Enrolled in another interventional research trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Barker, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Hospital, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arnsten AFT, Ishizawa Y, Xie Z. Scientific rationale for the use of alpha2A-adrenoceptor agonists in treating neuroinflammatory cognitive disorders. Mol Psychiatry. 2023 Nov;28(11):4540-4552. doi: 10.1038/s41380-023-02057-4. Epub 2023 Apr 7. PMID 37029295

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Guanfacine
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients admitted to surgical intensive care units at the University of Alabama at Birmingham Hospital.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Guanfacine | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 23 | 44
  >=65 years | 29 | 27 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.87 (13.95) | 65.36 (12.95) | 65.615 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 27 | 26 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 50 | 50 | 100
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 14 | 20
  White | 42 | 35 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100
Delirium Type [Number; unit: participants] — A positive Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) indicates delirium, while a negative result suggests its absence. Delirium subtypes were assigned by adding CAM-ICU with the Richmond Agitation-Sedation Score (RASS). Hypoactive delirium was diagnosed if CAM-ICU was positive and RASS score was -3 to 0, characterized by reduced activity and withdrawal. Hyperactive delirium was diagnosed if CAM-ICU was positive and RASS score was +1 to +4, associated with agitation and aggression. Mixed-type delirium occurred when both hypoactive and hyperactive symptoms were observed.
  participants
    Hypoactive Delirium | 36 | 40 | 76
    Hyperactive Delirium | 4 | 5 | 9
    Mixed Delirium | 10 | 4 | 14
    Coma | 0 | 1 | 1
APACHE II Score [Mean (Standard Deviation); unit: Score on a Scale] — APACHE II (Acute Physiology and Chronic Health Evaluation II) measures disease severity and predicts patient mortality. Age (0 to >75 years), temperature, mean arterial pressure, heart rate, respiratory rate, oxygenation, arterial pH, serum sodium, serum potassium, serum creatinine, hematocrit, white blood cell count, and Glasgow Coma Scale (scored 0 to 4 or 0 to 3), immunocompromised, hepatic failure, renal failure, hematologic malignancy, scored as none, mild, or severe (0 to 5 points). Score is a sum from 0 to 71, higher score indicates severe disease and worse outcome.
  Score on a Scale | 21.6 (6.4) | 21.1 (6.6) | 21.3 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Days Without Delirium
Description: The primary outcome will be the number of days alive without delirium during the 14-day treatment period after randomization. Delirium assessments are measured by the Confusion Assessment Method- Intensive Care Unit (CAM-ICU). CAM-ICU measures a patient's fluctuations in mental status, inattention, disorganized thinking, and consciousness.The CAM-ICU will be used twice daily with all patients while admitted until ICU discharge. Patients will be diagnosed as delirious when they have at least one positive CAM-ICU on the day of assessment up to ICU discharge or day 14 after enrollment if remaining in ICU. Patients will be diagnosed as delirium free when they have four (4) negative consecutive CAM-ICU assessments.
Time Frame: From the time of ICU admission up to 14 days
Population: Patients admitted to surgical intensive care unit at University of Alabama at Birmingham that received the study medication Guanfacine or Placebo.
Measure: Mean (Standard Deviation); unit: delirium free days
Arm/Group | Placebo | Guanfacine
Number analyzed (Participants) | 50 | 50
delirium free days | 2.54 (3.14) | 3.38 (3.70)
Statistical Analysis 1: Comparison: Placebo vs Guanfacine; Test type: Superiority; p = 0.22, t-test, 2 sided; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [2.3 to 4.4], Standard Deviation 3.7
Statistical Analysis 2: Comparison: Placebo vs Guanfacine; Null Hypothesis: The administration of guanfacine in critically ill patients in the intensive unit has no effect on the duration of delirium. Continuous variables will be summarized using sample mean and sample variance whereas categorical variables will be summarized as proportions. Logistic regression models will examine whether age, gender, or comorbities associated with incidence of delirium when Guanfacine is administered; Test type: Superiority; p = 0.0150, Regression, Linear — unadjusted for covariates; Risk Ratio (RR) = 1.3307, 95% CI 2-sided [1.0571 to 1.6751]

ADVERSE EVENTS:
Time Frame: 2 years, 6 months
Arm/Group | Placebo | Guanfacine
All-Cause Mortality (participants affected / at risk) | 10/50 | 9/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
This study is limited by the nature of being a single center design with a small sample size. The study population is in the critically ill surgical patient and this acuity and demographic may limit the external validity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT04578886/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT04578886/ICF_001.pdf